CLINICAL TRIAL: NCT01082523
Title: "A Randomized, Controlled, Evaluator-blinded Pilot Study to Evaluate the Effect of Automated Text Message Reminders on Patient Compliance With Topical Medications and Its Efficacy on Skin Disease Control in Adolescents and Adults With Mild to Moderate Acne"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2008-AB_01
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Acne; Patient Compliance
MeSH Terms: conditions — Acne Vulgaris; Patient Compliance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text message reminders (Active Comparator)
  Interventions: Other: Text message reminders
- Control (No Intervention)

INTERVENTIONS:
Other: Text message reminders — Subjects in this arm will receive twice daily automated text messages reminding them to apply their medications.
  Arms: Text message reminders

SUMMARY:
The purpose of this study is to determine whether an automated electronic reminder system using text messages sent to patient's cell phones will help patients with acne be more compliant with their topical medications and lead to an improvement of their acne.

Hypothesis: Automatically delivered electronic reminders in the form of text messages will increase acne patient adherence to topical medications and consequently result in better treatment outcome and higher patient satisfaction

DETAILED DESCRIPTION:
Patient non-compliance with topical medication use is a significant determinant of treatment failure resulting in both patient and physician frustration with outcome and leading to suboptimal medical care. It is important to address ways to improve patient compliance both from a medical and economic standpoint, as adequate use of medications could lead to a reduction of unnecessary office visits and a more cost-effective use of prescribed medications.

Patients with mild to moderate acne will be prescribed a standard treatment regimen with clindamycin/benzoyl peroxide gel in the mornings and adapalene gel in the evenings. Half of the subjects will then be randomly assigned to receive customized text messages instructing them twice a day to apply their morning and evening cream as prescribed, with the remainder of subjects serving as controls. Each medication tube supplied to every subject will be fitted with an electronic Medication Event Monitoring System cap (MEMS cap) which has the ability to record the date and time of every opening/closing of the tube. This data will serve as an objective measure of medication use and will be used to determine whether the reminder messages resulted in a higher and more consistent use of the prescribed medications.

Specific Aims:

The primary aim of the study is to determine whether automated text messages produce increased adherence with medication use in the Reminder group compared to the Control group over the 12 week study duration.

Improvement in acne will be measured using full face lesion counts, Investigator Global Assessment Score (IGA) and subject Global Assessment Score (SGA). Quality of life and satisfaction will be measured using the Dermatology Life Quality Index (DLQI), and patient satisfaction surveys.

ELIGIBILITY:
Inclusion Criteria:

* males and females 12-30 years of age at time of consent
* any ethnic background
* be capable of giving informed consent
* have clinical diagnosis of acne vulgaris with facial involvement for at least 6 months prior to enrollment.
* Must have a minimum of 30 to 100 non-inflammatory facial lesions (open and/or closed comedones), and 20 to 50 inflammatory lesions (papules or pustules) and no nodules or cysts.
* Must have a score 2 or 3 on the Investigator Global Assessment Scale (IGA)
* Must own a personal mobile telephone with SMS text messaging capabilities.
* Must be English or Spanish speaking.
* Women of child bearing potential and all men must be using adequate birth control measures (e.g. abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) and must agree to continue to use such measures and not become pregnant or plan a pregnancy until 12 months after receiving the last dose of study medication.
* Must be able to adhere to study visit schedule and other protocol requirements.
* Must avoid prolonged sun exposure and avoid use of tanning booths or other ultraviolet light sources during the study.
* Must agree not to use any other prescription or over the counter medications other than the ones prescribed by the study protocol.
* Must agree to limit Vitamin A supplementation to total daily dose 4000-5000 IU.

Exclusion Criteria:

* Nodular or cystic acne, acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced, mechanical)
* Known exposure history to environmental or chemical comedogenic agents such as cutting oils, tar, halogenated compounds or polyaromatic hydrocarbons.
* Women with a known history or clinical evidence of hyperandrogenism such as polycystic ovarian syndrome.
* Known history or clinical evidence of Cushing's syndrome or congenital adrenal hyperplasia.
* Use of hormonal contraceptives or intrauterine device (unless subject is on stable dose, i.e at least 6 months of prior treatment
* Have used any investigational drug within the previous 4 weeks or 5 times the half life of the investigational drug, whichever longer.
* Have received phototherapy or use a tanning booth within 4 weeks prior to enrollment
* Currently taking any systemic medications that could affect evaluation of acne (including, but not limited to antibiotics, retinoids, biologic disease modifying agents, chemotherapeutic agents, anti-epileptic agents or EGFR-receptor antagonists)
* History of chronic or recurrent infectious disease, including, but not limited to folliculitis, infected skin wounds or ulcers and recurrent herpes simplex infections.
* Known hypersensitivity response, including anaphylaxis, to any of the compounds used for treatment (e.g: clindamycin, retinoids).
* Known substance abuse (drug or alcohol) problem within the previous 12 months.
* Presence of beard or facial hair which might interfere with study assessments
* Participating in another clinical trial using an investigational agent or procedure during participation in the study.
* Are pregnant or planning pregnancy or a surgery during the participation in the study

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
adherence to topical medication use | 12 weeks
  The primary goal of the study is to determine whether automated text messages produce increased adherence with medication use in the Reminder group compared to the Control group over the 12 week study duration. Overall adherence will be calculated as the total number of doses applied (recorded cap opening/closing events) divided by the total number of expected doses applied (twice daily cap opening/closing events) based on the prescribed treatment regimen.

SECONDARY OUTCOMES:
Improvement in acne severity (as measured by IGA score) | 12 weeks
  Secondary endpoints include determination of improvement in acne severity, quality of life, and patient satisfaction in the Reminder versus Control group at study completion (week 12 compared to baseline). Improvement in acne will be measured using full-face lesion counts, Investigator Global Assessment Score (IGA) and subject Global Assessment Score (SGA). Quality of life and satisfaction will be measured using the Acne Quality Index Index(Acne-QoL), and patient satisfaction surveys.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UT Southwestern Medical Center at Dallas - Dermatology Clinical Trials, Dallas, Texas
  - Department of Dermatology, University of Texas Southwestern Medical Center, Dallas, Texas